CLINICAL TRIAL: NCT02782312
Title: Salmeterol-Fluticasone Combined Inhaled Therapy for Non-cystic Fibrosis Bronchiectasis With Airway Limitation: a Prospective Study
Brief Title: Salmeterol-Fluticasone Combined Inhaled Therapy for Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director of respiratory department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110505
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; ICS+LABA
MeSH Terms: conditions — Bronchiectasis | interventions — Fluticasone-Salmeterol Drug Combination

ARMS (2):
- ICS+LABA Group (Experimental): Seretide 250，inhalation，twice daily，one year
  Interventions: Drug: ICS+LABA
- Control Group (Active Comparator): routine therapy for one year
  Interventions: Other: routine therapy

INTERVENTIONS:
Drug: ICS+LABA — Seretide is inhaled for one year
  Other Names: Seretide
  Arms: ICS+LABA Group
Other: routine therapy — routine therapy for one year
  Arms: Control Group

SUMMARY:
The objective of this study is to assess the efficacy and safety of Salmeterol-Fluticasone （ICS and LABA）combined inhaled therapy for non-cystic fibrosis（non-CF）bronchiectasis patients with chronic airflow obstruction. Moreover, subgroup analysis is performed to explore which populations of bronchiectasis patients this treatment is suitable for.

DETAILED DESCRIPTION:
Inhaled ICS and LABA have proved obvious benefit for asthma or chronic obstructive pulmonary disease (COPD) patients. However, there is presently no clear evidence on the effect of ICS and LABA combined inhaled therapy for non-CF bronchiectasis patients.

This study is designed as a prospective, randomized,control trial. Patients are divided into two groups, one group inhaled with ICS and LABA (Seretide), another group received routine therapy (oxygen uptake, phlegm dissipation, hemostasis postural drainage and naturopathy).The course of treatment is 12 months. All patients underwent reviews at baseline entry to the study and at months 6 and 12 of treatment.

The quality of life (QOL) scores：St George's dyspnea score (SGRQ score）, modified british medical reserach council（mMRC score) and COPD assessment test (CAT score); lung function test: forced expiratory volume in one second (FEV1）,FEV1% predicted, the ratio of forced expiratory volume in one second and forced vital capacity (FEV1/FVC%); short-acting β2-adrenergic agonist（SABA）use and the incidence of adverse event were monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* stable bronchiectasis; have the ability to complete the pulmonary function tests; FEV1/FVC<70%; ≥2 exacerbations within the past year

Exclusion Criteria:

* a cigarette smoking history more than 10 pack-years;cystic fibrosis or traction bronchiectasis due to various pulmonary fibrosis; an active pulmonary mycobacterial infection; fungal infection; active sarcoidosis; active allergic bronchopulmonary aspergillosis (ABPA); asthma as defined by the Global Initiative for Asthma (GINA); patients with severe cardiopulmonary dysfunction; with impaired hepatic or kidney function; with hypogammaglobulinemia or other autoimmune diseases; pregnant or breast-feeding women; or patients with a known intolerance for ICS or LABAs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 months
  CAT score
Quality of life | 12 months
  mMRC score
Quality of life | 12 months
  SGRQ score

SECONDARY OUTCOMES:
pulmonary function text | 12 months
  FEV1
pulmonary function text | 12 months
  FEV1% predicted
pulmonary function text | 12 months
  FEV1/FVC
short-acting β2-adrenergic agonist (SABA) used | 12 months
  Number of SABA needed per patient every week
Exacerbations | 12 months
  The times of acute exacerbation during the trial.
sputum microorganism culture | 12 months
  Number of microorganism isolates along the study
Number of patients with adverse events | 12 months
  All of the adverse events occurred in the processing of the trial,especially adverse events associated with inhaled corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, Principal Investigator — Shanghai Pulmonary Hospital , Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Martinez-Garcia MA, Soler-Cataluna JJ, Catalan-Serra P, Roman-Sanchez P, Tordera MP. Clinical efficacy and safety of budesonide-formoterol in non-cystic fibrosis bronchiectasis. Chest. 2012 Feb;141(2):461-468. doi: 10.1378/chest.11-0180. Epub 2011 Jul 21. PMID 21778259
- [Result] Tsang KW, Tan KC, Ho PL, Ooi GC, Ho JC, Mak J, Tipoe GL, Ko C, Yan C, Lam WK, Chan-Yeung M. Inhaled fluticasone in bronchiectasis: a 12 month study. Thorax. 2005 Mar;60(3):239-43. doi: 10.1136/thx.2002.003236. PMID 15741443
- [Result] Goyal V, Chang AB. Combination inhaled corticosteroids and long-acting beta2-agonists for children and adults with bronchiectasis. Cochrane Database Syst Rev. 2014 Jun 10;2014(6):CD010327. doi: 10.1002/14651858.CD010327.pub2. PMID 24913725